CLINICAL TRIAL: NCT03202485
Title: Comparison Between Toric and Spherical Implantable Collamer Lens Combined With Astigmatic Keratotomy for High Myopic Astigmatism
Brief Title: Comparison Between TICL and ICL+AK for High Myopic Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, vice director of refractive surgery department of the eye hospital of WZMU, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TICL compare with ICL+AK
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Astigmatism; High Myopia
Keywords: astigmatism; high myopia; phakic intraocular lens; astigmatic keratotomy; toric
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective comparative case series
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric Implantable Collamer Lens (Active Comparator): Subjects in this group will implant Toric Implantable Collamer Lens for high myopic astigmatism
  Interventions: Device: Toric Implantable Collamer Lens
- ICL+ Astigmatic keratotomy (Experimental): Subjects in this group will implant Implantable Collamer Lens and combined with astigmatic keratotomy for high myopic astigmatism
  Interventions: Device: ICL + Astigmatic keratotomy

INTERVENTIONS:
Device: Toric Implantable Collamer Lens — uses Toric Implantable Collamer Lens implantation to correct the high myopic astigmatism.
  Arms: Toric Implantable Collamer Lens
Device: ICL + Astigmatic keratotomy — uses Implantable Collamer Lens implantation combined with Astigmatic keratotomy to correct the high myopic astigmatism
  Arms: ICL+ Astigmatic keratotomy

SUMMARY:
To compare the outcomes of a toric Implantable Collamer Lens (ICL) and a spherical Implantable Collamer Lens combined with astigmatic keratotomy (AK) in the correction of high myopic astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 18 to 40 years,
* myopia greater than -8.00 diopters (D), and refractive cylinder in the range of 1.50D to 5.50D,
* for the patients who were planned to undergo AK+ICL implantation, the axial difference between the corneal astigmatism and the manifest refractive astigmatism was less than 10 degree,
* a stable refractive error during the previous 2 years,
* anterior chamber depth more than 2.8 mm,
* endothelial cell density (ECD) more than 2500 cells/mm2, and
* scotopic pupillary diameter less than 7 mm.

Exclusion Criteria:

* subjects had significant irregular astigmatism, corneal pathological changes, glaucoma, ocular inflammation, or previous ocular trauma or surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity (UCVA) at distance | 2 years after surgery
  measured at 5 meter
astigmatism | 2 years after surgery
  astigmatism getting from subjective refraction

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) at distance | 2 years after surgery
  subjective refraction
Spherical Equivalent (SE) | 2 years after surgery
  subjective refraction
mean postoperative BCVA/mean preoperative BCVA | 2 years after surgery
  safety index
mean postoperative UCVA/mean preoperative BCVA | 2 years after surgery
  efficacy index

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD.PhD., Principal Investigator — Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng LY, Zhu SQ, Su YF, Zou HY, Wang QM, Yu AY. Comparison between toric and spherical phakic intraocular lenses combined with astigmatic keratotomy for high myopic astigmatism. Eye Vis (Lond). 2017 Aug 18;4:20. doi: 10.1186/s40662-017-0085-7. eCollection 2017. PMID 28828390